CLINICAL TRIAL: NCT03358173
Title: Operative Plate Fixation Versus Conservative Treatment for Acute, Displaced Fractures of Humeral Shaft
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, pengzhang, Department of orthopaedics and trauma, Peking University People's Hospital
Other Study IDs: csg-ggggz
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Humeral Fractures
Keywords: Humeral Fractures; plate; Conservative Treatment
MeSH Terms: conditions — Humeral Fractures | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conservative Treatment: Standard protocol for conservative treatment will consist of the implementation of a sling and patient comfort. Pendulum or gentle Range of Motion (ROM) shoulder exercises may be implemented at any time as dictated by the attending surgeon.
  Interventions: Procedure: Conservative Treatment
- Operative Plate Fixation: The operating surgeon will determine the positioning of the patient for surgery. ORIF of the humeral shaft fracture will be carried out
  Interventions: Procedure: Operative Plate Fixation

INTERVENTIONS:
Procedure: Conservative Treatment — Conservative Treatment
  Groups: Conservative Treatment
Procedure: Operative Plate Fixation — Operative Plate Fixation
  Groups: Operative Plate Fixation

SUMMARY:
Conservative Treatment Versus Operative Plate Fixation for Acute, Displaced Fractures of the Distal Clavicle

DETAILED DESCRIPTION:
From Jane 2015 to October 2016, patients with displaced humeral shaft fractures are retrospectively included in this study, they were treated with either operative plate or conservative treatment. All the patients are regularly followed up in clinic. Then we will compare the union rate and clinical functional outcome(DASH score) between the 2 groups at 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

Men or women aged 18 to 65 years of age Completely displaced ,closed fracture of humeral shaft confirmed by radiograph Fractures within 1 month post injury Provision of informed consent

Exclusion Criteria:

Pathological fractures Non-displaced (cortical contact) fractures Open fractures Presence of vascular or nerve injury Fractures more than 1 month post-injury Limited life expectancy due to significant medical co-morbidity Medical contraindication to surgery Inability to comply with rehabilitation or form completion Likely problems, in the judgement of the investigators, with maintaining follow-up (i.e. patients with no fixed address, patients not mentally competent to give consent, etc.)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men or women aged 18 to 65 years of age Completely displaced ,closed fracture of humeral shaft confirmed by radiograph Fractures within 1 month post injury
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2017-12-25 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Union rate | 1 year after surgery
  Union rate of the fracture from X-ray

SECONDARY OUTCOMES:
Functional score | 1 year after surgery
  DASH score of the injured arm

CONTACTS AND LOCATIONS:
Overall Officials: Peng Zhang, MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No